CLINICAL TRIAL: NCT05368389
Title: Observational Feasibility Study of the Healthdot Wearable Monitoring Device in Bariatric Patients at Mayo Clinic
Brief Title: Observational Study of Wearable Health Monitoring Device
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: Philips Healthcare (Industry)
Responsible Party: Principal Investigator, Eric J. Vargas Valls, Principal Investigator, Mayo Clinic
Other Study IDs: 21-007489
Record Dates: First submitted 2022-05-06; First posted 2022-05-10 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Weight Loss
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- Healthdot Patients: This group represents the patient who have undergone a bariatric procedure and had the Healthdot device attached and had data collected from the device for 10 days.
  Interventions: Device: Healthdot attachment
- Healthdot providers: This group represents the providers or study/hospital staff who were involved in the attachment, recruitment, and enrollment of the Healthdot patients.

INTERVENTIONS:
Device: Healthdot attachment — The wearable health monitoring device "Healthdot 5" will be attached to the patient's skin at left lower rib and data like heart rate, respiratory rate, posture and activity will be collected for 10 days.
  A questionnaire will be sent to patients to fill out at the 10th day after the device attachment.
  Groups: Healthdot Patients

SUMMARY:
The purpose of this study is to better understand the use of Healthdot devices on bariatric patients in the USA. Healthdot is a wearable monitoring device that can collect data on heart rate, respiration rate, posture, and activity. This device can be worn at the hospital and at home. The Healthdot will be able to send data and have good connectivity in a place where there is network coverage(4G/5G).

DETAILED DESCRIPTION:
This clinical study is a single-center observational feasibility study of the Healthdot device, a wearable health monitoring device applied to bariatric surgery/endoscopy patients for in-hospital and at-home data collection of heart rate, respiration rate, posture, and activity. After surgery, 30 bariatric patients will be applied with the Healthdot device. Patient data will be collected for a total of 10 days to evaluate the feasibility of the use of the Healthdot device at Mayo Clinic and at home. Patient data will only be observed retrospectively, so after the data collection period of 10 days has been concluded, the clinical care will not be affected by this. Feasibility includes the connectivity performance, the usability from a hospital staff perspective with a focus on staff satisfaction and potential interference with hospital workflow, and the usability from a patient perspective with a focus on patient satisfaction and potential interference with normal daily activities. The collected information will be processed to establish the feasibility of a larger interventional clinical trial using Healthdot in bariatric patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients being seen for upcoming planned weight-loss procedure (ESG, Balloon, Bariatric Surgery, Revision after Bariatric Surgery).
* Commitment to wear device without removing for entire study period.
* Located within a driving distance from Mayo Clinic in Rochester, Minnesota during study duration.
* Reside in an area with 4G or 5G connectivity based on cellphone provider maps for T-Mobile or AT&T.
* Subject clear of any dermatologic health diagnosis that may impede the ability of the device to adhere properly.

Exclusion Criteria:

* Unable to give consent.
* Unwillingness to utilize email address for device instructions, surveys, and reminders.
* Lifestyle that would have the device exposed to excessive elements for a prolonged period of time outside the parameters of normal operation of the device.
* Patient is expected/anticipated to fly (use an airplane) before study completion (before Day 10).
* Subjects with a pacemaker or an implanted electronic device.
* Subjects scheduled or likely to conduct MRI within the study period.
* Left lower rib (place where Healthdot will be applied) is involved in the area of surgery, area of disinfection or area where bandages are needed.
* Patients with severe systemic diseases.

Ages: 22 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: In this clinical study, 30 patients undergoing a bariatric procedure (ESG, Balloon, Bariatric Surgery, Revision after Bariatric Surgery) will be enrolled.
  An estimate of 10 providers/Hospital Staff will be accrued for the study to fill out a provider satisfaction questionnaire regarding the Healthdot device.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2022-11-03 (Actual); Primary Completion 2023-06-21 (Actual); Study Completion 2023-06-21 (Actual)

PRIMARY OUTCOMES:
Transmit number | 10 days
  The number of times data is collected successfully from the Healthdot device.

SECONDARY OUTCOMES:
Patient Satisfaction Questionnaire | Day 10
  The questionnaire will be sent to bariatric patients with questions regarding the usability and satisfaction wearing the healthdot device. The answer will be represented in multiple choices. The answers will be collected and the data will be analyzed.
  Each question will be scored on a likert scale 0 being the lowest score and 5 the highest.
Provider Satisfaction Questionnaire | 6 month
  The questionnaire will be sent to providers and Study staff with questions regarding the usability and satisfaction of using and attaching the Healthdot device in the hospital setting. The answer will be represented in multiple choices and open answers. The answers will be collected and the data will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Eric K Vargas Valls, MD, MS, Principal Investigator — Mayo Clinic
Locations (1):
- Karl Akiki, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials/cls-20537138